CLINICAL TRIAL: NCT04622930
Title: Smartphone Cognitive Behavioral Therapy for Social Anxiety Disorder: A Randomized, Waitlist-control Trial
Brief Title: Waitlist-Control Trial of Smartphone (App-based) CBT for Social Anxiety Disorder (SAD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer proceeding with this study.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Koa Health B.V. (Industry)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Chief of Phycology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001671; NCT03769363 (obsolete NCT alias)
Record Dates: First submitted 2020-10-13; First posted 2020-11-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Sagittal Abdominal Diameter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental: Smartphone-delivered CBT for SAD (Experimental): 12-week Smartphone delivered CBT for SAD.
  Interventions: Device: Smartphone-delivered CBT for SAD
- 12 Week Waitlist Control (Other): 12-week waitlist control. (Note: participants will be crossed over to 12-week Smartphone-delivered CBT for SAD following the 12-week waitlist control).
  Interventions: Device: Smartphone-delivered CBT for SAD

INTERVENTIONS:
Device: Smartphone-delivered CBT for SAD — 12-week Smartphone-delivered CBT for SAD. In-person cognitive-behavioral therapy (CBT) is an empirically supported treatment for SAD. The app-delivered CBT in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work), behavioral skills (e.g., exposure with ritual prevention), and perceptual retraining/mindfulness skills.

SUMMARY:
The investigators are testing the efficacy of Smartphone-delivered cognitive behavioral therapy (CBT) treatment for social anxiety disorder (SAD). The investigators hypothesize that participants receiving app-CBT will have greater reduction in LSAS scores than those in the waitlist condition at treatment endpoint (week 12).

DETAILED DESCRIPTION:
The primary aims of this study are to test the efficacy of a Smartphone-based CBT treatment for adults with SAD recruited nationally. Eligible subjects (N=80) will be randomly assigned to 12 weeks of Smartphone-delivered CBT for SAD either immediately, or after a 12-week long waiting period (50-50 chance). The investigators hypothesize that Smartphone-delivered CBT for SAD will be feasible and acceptable to individuals with SAD, and that it will lead to greater reductions in SAD symptom severity compared to the passage of time (waitlist control).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Current diagnosis of primary DSM-5 SAD, based on MINI
* Currently living in the United States

Exclusion Criteria:

* Psychotropic medication changes within 2 months prior to enrollment i. Participants taking psychotropic medication must have been on a stable dose for at least 2 months prior to enrollment and not change medication during study period
* Past participation in ≥ 4 sessions of CBT for SAD
* Current severe substance use disorder
* Lifetime bipolar disorder or psychosis
* Current severe comorbid major depression, as indicated by clinical judgment and/or a QIDS-SR total score ≥ 21 ***EDIT***
* Acute, active suicidal ideation as indicated by clinical judgment and/or a score ≥ 2 on the suicidal ideation subscale of the C-SSRS
* Concurrent psychological treatment
* Does not own a supported mobile Smartphone with a data plan
* Lack of technology literacy that would interfere with ability to engage with smartphone treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in SAD severity (LSAS) at the end of treatment/waitlist period. | Endpoint (week 12)
  The Liebowitz Social Anxiety Scale (LSAS) is a clinician-administered measure of social anxiety symptom severity. It contains 24 social situations likely to elicit social anxiety, and items are scored on a Likert scale ranging from 0 to 3. Higher scores indicate more severe SAD symptoms. The LSAS will be used to assess change in social anxiety symptoms from baseline to endpoint.

SECONDARY OUTCOMES:
Difference in depression severity as assessed by change in The Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) total scores from baseline to week 12. | Endpoint (week 12)
  Participants who receive app-CBT will have a difference in depression severity as assessed by change in The Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) total scores from baseline to week 12. The CESD-R is a self-report measure of depressive symptoms consisting of 20 scale items with responses ranging from 0 to 4, including two questions about suicidal ideation (item #14, #15). Higher scores correspond with greater depression severity, and the measure is a well-validated, sensitive measure of symptom severity in depression.
Difference in functional impairment as measured by change in The Work and Social Adjustment Scale (WSAS) total scores from baseline to week 12. | Endpoint (week 12)
  Participants who receive app-CBT will have a difference in functional impairment as measured by change in The Work and Social Adjustment Scale (WSAS) total scores from baseline to week 12. The WSAS uses a Likert scale from 0 (not at all impaired) to 8 (very severely impaired) to assess impairment in occupational, social, and family/friends domains. Higher scores indicate greater impairment.
Difference in quality of life as assessed by change in The Quality of Life, Enjoyment, and Satisfaction Questionnaire-Short Form (QLESQ-SR) total scores from baseline to week 12. | Endpoint (week 12)
  Participants who receive app-CBT will have a difference in quality of life as assessed by change in The Quality of Life, Enjoyment, and Satisfaction Questionnaire-Short Form (QLESQ-SR) total scores from baseline to week 12. The Q-LES-Q-SF is a self-report measure of subjective quality of life, containing Likert items ranging from 1 (Very Poor) to 5 (Very Good). Total scores are presented as a percentage of the maximum value (i.e., ranging from 0 to 100, with higher scores indicating greater quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States